CLINICAL TRIAL: NCT02567383
Title: A Phase II Clinical Trial Evaluating the Safety and Efficacy of Combination of Hyperthermia and Concurrent Chemoradiotherapy (CCRT) for Recurrent Head and Neck Cancer
Brief Title: Combination of Hyperthermia and Concurrent Chemoradiotherapy (CCRT) for Recurrent Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150205D
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Head and Neck Cancer
Keywords: head and neck cancer; hyperthermia, Thermotron RF-8; radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Hyperthermia | interventions — Radiation; Diathermy; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperthermia (Experimental): Hyperthermia; Thermotron RF-8, radiation, Cisplatin and Taxotere
  Interventions: Radiation: Radiation; Device: Hyperthermia; Thermotron RF-8; Drug: Cisplatin; Drug: Taxotere

INTERVENTIONS:
Radiation: Radiation — 5-Gy once a week for a subtotal of 10Gy/2fx a week to gross tumors, followed by 40Gy/20fx/4 weeks, total 50Gy/22fx/5weeks
Device: Hyperthermia; Thermotron RF-8 — 40 minutes within 2hr after irradiation
Drug: Cisplatin — 20mg/m2 per week for 6 weekly cycles before radiotherapy
Drug: Taxotere — 10-12mg/m2 per week for 6 weekly cycles before radiotherapy

SUMMARY:
Clinical experience of with hyperthermia combined with radiotherapy and chemotherapy for recurrent head and neck cancer is limited. The primary goals of hyperthermia combined with CCRT on recurrent head and neck cancer are tumor response rate, while secondary goals are rates of acute and late adverse effects, local control rate, distant metastasis rate, progression-free rate and overall survival rate.

DETAILED DESCRIPTION:
Patients will be treated with radiotherapy with 50Gy/22fx/6 weeks, plus hyperthermia for 40 minutes within 2hr after irradiation, with maximum temperature setted on 42℃ ± 0.5℃ as upper limit, once a week since the 1st week of radiation for a total of 6 times. The regimen of concurrent chemotherapy will be cisplatin 20mg/m2 and taxotere 10-12mg/m2 per week for 6 weekly cycles on the day before radiotherapy and hyperthermia treatment. The two chemotherapy agents will be given in only one day every week, according to the weekly dose. According to Gehan two-stage design, provided the estimated tumor response rate using this regimen is about 40% and objective tumor response is observed in ≥1 of the first 6 patients enrolled, α<0.05 will be achieved indicating a preliminary efficacy. Then the Gehan second stage will be started. With a set of 5% precision and an assumption of 10% dropout rate, 39 additional patients will be enrolled in the Gehan second stage depending on the actual number with tumor response in the Gehan first stage (totaling 45 patients when counting the first 6 in the Gehan first stage). The tumor response, adverse effects and various survival curves will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20-85 years, with ECOG performance 0-2.
2. Treatment failure head and neck cancer, with histologically or clinically confirmed recurrence or progression after previous treatment of radiotherapy with combinations.
3. Complete surgical excision is NOT feasible as salvage treatment for the recurrent or progressive tumor(s), or the patient does NOT agree to receive the surgical procedure.
4. Salvage radiotherapy is possible, and a total dose of 50Gy/22fx is considered tolerable.
5. Measurable lesions by image examinations or endoscopy within 2 months.
6. The distribution of the lesions of interest does NOT exceed 20cm range.
7. The patient can tolerate implementation of cisplatin and taxotere weekly therapy, with respect to hematopoietic status, renal function, liver function, allergy and other potential adverse effects.
8. There is NO other effective treatment option according to the evaluation of physicians.

Exclusion Criteria:

1. Re-irradiation of 50Gy/22fx is considered NOT tolerable.
2. Future tumor response to treatment in this study is NOT possibly evaluated using image examinations or endoscopy.
3. The patient is participating in other clinical trials.
4. Future regular clinical follow-up is NOT possible.
5. The patient has large-area metallic implants or tattoos including much metal powder within hyperthermia field (not including metallic hemoclips with small area and few numbers).
6. The patient has pacemakers, electrocardiograph, defibrillator implanted, or adhesive skin patches including conductive metal.
7. The patients with ocular or cerebral disorders within hyperthermia field.
8. Tumor invasion of great or large vessels exists, or patients with any existing complications that may pose risks to hyperthermia treatment.
9. Patients who have difficulty with communication.
10. Other patients who are considered to have a contraindication to hyperthermia treatment.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | 12 Weeks
  To estimate the tumor response rate (complete response + partial response; CR + PR; according to RECIST criteria version 1.1) using hyperthermia combined with CCRT for recurrent head and neck cancer.

SECONDARY OUTCOMES:
Adverse events | Within 3 months
  To estimate rates of each grade adverse events (CTCAE, version 4.0) which is possibly, probably, or definitely related to treatment and which occurs within 3 months from the start of radiation combined with hyperthermia and chemotherapy.
Late adverse events | After 3 months
  To estimate rates of late adverse events (3 months from start of radiation combined with hyperthermia and chemotherapy)

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang KL, Chi MS, Hao CY, Ko HL, Huang YY, Wu RH, Lai HC, Lin YC, Hao SP, Chi KH. Phase II clinical trial assessing the addition of hyperthermia to salvage concurrent chemoradiotherapy for unresectable recurrent head and neck cancer in previously irradiated patients. Radiat Oncol. 2025 Feb 8;20(1):21. doi: 10.1186/s13014-025-02585-z. PMID 39920700